CLINICAL TRIAL: NCT07054190
Title: A Phase II, Open-Label, Multicenter Study Evaluating the Safety and Efficacy of Neoadjuvant Treatment With Inavolisib Combinations in Patients With Untreated, Early-stage, PIK3CA-Mutated Breast Cancer
Brief Title: A Study to Test Inavolisib Treatments in Participants With Early-Stage, PIK3CA-Mutated Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO45853; 2024-518811-20-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — inavolisib; ribociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Participants will receive inavolisib and letrozole orally (PO) once a day (QD) from Day 1 to 28 and ribociclib PO QD from Day 1 to 21 in cycles 1-5 (each cycle=28 days). In cycle 6, inavolisib, ribociclib and letrozole will be administered PO QD on days 1-21 (each cycle=21 days).
  Interventions: Drug: Inavolisib; Drug: Ribociclib; Drug: Letrozole
- Arm B (Experimental): Participants will receive a starting regimen of inavolisib and letrozole PO QD from Day 1 to 28 in cycle 1 (each cycle=28 days). Starting on Day 1 of Cycle 2, all participants will receive the triplet regimen inavolisib + ribociclib + letrozole as follows: inavolisib and letrozole PO QD from Day 1 to 28 and ribociclib PO QD from Day 1 to 21 in cycles 2-5 (each cycle=28 days). In cycle 6, inavolisib, ribociclib and letrozole will be administered PO QD on days 1-21 (each cycle=21 days).
  Interventions: Drug: Inavolisib; Drug: Ribociclib; Drug: Letrozole
- Arm C (Experimental): Participants will receive a starting regimen of ribociclib PO QD from Day 1 to 21 and letrozole PO QD from Day 1 to 28 in cycle 1 (each cycle=28 days). Starting on Day 1 of Cycle 2, all participants will receive the triplet regimen inavolisib + ribociclib + letrozole as follows: inavolisib and letrozole PO QD from Day 1 to 28 and ribociclib PO QD from Day 1 to 21 in cycles 2-5 (each cycle=28 days). In cycle 6, inavolisib, ribociclib and letrozole will be administered PO QD on days 1-21 (each cycle=21 days).
  Interventions: Drug: Inavolisib; Drug: Ribociclib; Drug: Letrozole

INTERVENTIONS:
Drug: Inavolisib — Inavolisib will be administered as per the schedule specified in the arms
  Other Names: GDC-0077; RO7113755
Drug: Ribociclib — Ribociclib will be administered as per the schedule specified in the arms
Drug: Letrozole — Letrozole will be administered as per the schedule specified in the arms

SUMMARY:
This study will evaluate the safety and efficacy of inavolisib combination therapies in participants with untreated, PIK3CA-mutated, Stage II-III, estrogen receptor (ER)-positive, Human Epidermal Growth Factor Receptor 2 (HER2)-negative breast cancer (BC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed operable or inoperable invasive Stage II-III BC according to American Joint Committee on Cancer (AJCC) TNM staging classification
* Candidate for neoadjuvant treatment and considered appropriate for endocrine combination therapy
* Willingness to undergo breast surgery (mastectomy or breast-conserving surgery) after neoadjuvant treatment (unless inoperable)
* Documented ER-positive tumor in accordance with current American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines
* Documented HER2-negative tumor in accordance with current ASCO/CAP guidelines
* Documented Ki-67 score >=5% as per local assessment
* Confirmed PIK3CA mutation

Exclusion Criteria:

* Stage IV (metastatic) BC
* Inflammatory BC (cT4d)
* Bilateral invasive BC
* History of ductal carcinoma in situ or lobular carcinoma in situ if they have received any systemic therapy for treatment or radiation therapy to the ipsilateral breast
* Previous systemic or local treatment for the primary BC currently under investigation (including excisional biopsy or any other surgery of the primary tumor and/or axillary lymph nodes, including sentinel lymph node biopsy, radiotherapy, cytotoxic, and endocrine treatments)
* Type 2 diabetes requiring ongoing systemic treatment at the time of study entry; or any history of Type 1 diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | From first dose up to 30 days after last dose (approximately 8 months)

SECONDARY OUTCOMES:
Percentage of Participants with Total Pathological Complete Response (pCR) | Up to approximately 8 months
Percentage of Participants with Objective Response Rate (ORR), According to Modified Response Evaluation Criteria in Solid Tumors, Version 1.1 (mRECIST v1.1) | Up to approximately 8 months
Change From Baseline in Ki-67 Levels by Immunohistochemistry (IHC) | Baseline, Day 22 of Cycle 1 and at Surgery (up to approximately 8 months). One cycle = 28 days
Percentage of Participants Reporting Symptoms in Patient-Reported Outcomes of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Questionnaire | Up to approximately 8 months
Percentage of Participants Reporting Each Response Option at Each Time Point for the Treatment Side-Effect Bother Item (GP5) From the Functional Assessment of Cancer Therapy - General (FACT-G) Questionnaire | Up to approximately 8 months
Change from Baseline in Symptomatic Treatment-Related Toxicities as Assessed Through use of the PRO-CTCAE | Baseline, up to approximately 8 months
Change from Baseline in Treatment Side-Effect Bother as Assessed Through use of the FACT-G GP5 Item | Baseline, up to approximately 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- Centro Oncologico Korben, Ciudad Autonoma Buenos Aires, Argentina
- Brazil (4):
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
- Canada (3):
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
- Germany (2):
  - Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Heidelberg, Heidelberg
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center., Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing